CLINICAL TRIAL: NCT02555969
Title: Minimal Residual Disease as a Possible Predictive Factor for Relapse in Patients With AL Amyloidosis
Status: Completed | Type: Observational
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 11829
Record Dates: First submitted 2015-09-16; First posted 2015-09-22 (Estimated); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Amyloidosis; Primary Amyloidosis
MeSH Terms: conditions — Amyloidosis; Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This protocol will assess patients with AL amyloidosis who achieve a complete response (CR) or very good partial response (VGPR) to therapy for minimal residual disease (MRD). Three approaches to MRD testing will be used since there is no established method. The investigators will clone and sequence each patient's light chain (LC) gene and design patient-specific primers to evaluate genomic DNA from future marrow specimens. Whole genome sequencing (WGS) will be used to test baseline and follow-up marrow cell DNA, seeking copy number variations in chromosomes 1 and 2 or 22, and structural variations in chromosomes 11 and 14, consistent with the known genetic abnormalities in AL and with clonal LC gene use. Plasma protein analysis by mass spectrometry will also be used to look for fragmentary protein sequences associated with the culprit LC gene of each subject. The feasibility and predictive value of these three approaches in patients achieving CR or VGPR will be evaluated. This protocol will help provide insight into the ways that the disease changes and progresses. MRD testing is likely an important next step in AL management.

DETAILED DESCRIPTION:
This protocol will assess AL amyloidosis patients who achieve a CR or VGPR to first-line therapy for evidence of MRD by Q-PCR, NGS, and plasma protein analysis by mass spectrometry using marrow cells obtained annually at times of standard clinical evaluations.

A bone marrow aspirate sample from diagnosis will be used to create a baseline profile of each patient's disease. This sample will allow the investigators to create the primer-probe sets required for MRD testing by Q-PCR, which will be conducted after the patient has achieved a CR or VGPR. A baseline bone marrow biopsy sample will either be taken at the time of consent or can be taken from storage if the patient has previously consented to have their marrow cells banked for research purposes. An extra 15 mL of aspirate will be taken from their diagnostic bone marrow biopsy, which is routinely conducted on newly diagnosed patients for clinical purposes. Annual bone marrow aspirates will not be taken for research purposes until after the patient has responded. Patients will remain on protocol, but only begin MRD testing after achieving a CR or VGPR to first-line therapy at which point annual marrow collections for MRD testing will begin. In the event the patient does not reach a CR or VGPR to first-line therapy, the baseline bone marrow aspirate from diagnosis will be discarded.

Patients who choose to allow their marrow to be used in this study will sign a consent form specifically for this study. At the time of consent, three green top tubes of peripheral blood will be obtained for WGS of non-tumor cells. No further blood samples will be required for this study. After achieving a CR or VGPR, patients will be completely re-staged as is standard of care at annual intervals. Samples to test for the presence of MRD in their marrows will be obtained at these times of clinical re-staging for up to 3 years after their response to therapy. Both blood and bone marrow samples for this study will be immediately taken to an on-site laboratory where they will be briefly stored before testing. This will ensure no study samples interfere with routine clinical care.

In order to test for the presence of MRD, three techniques will be used: Q-PCR, WGS, and plasma protein analysis by mass spectrometry. Both Q-PCR and WGS will use genomic DNA from marrow aspirate samples. To make primer-probe sets for Q-PCR, bone marrow samples from baseline will be used to create individualized primer-probe sets that can recognize the genetically unique LC gene that causes each patient's disease. To perform WGS, genomic DNA will be supplied to the core genetics laboratory for creation of a library and multiplex next generation sequencing. To perform plasma protein analysis, plasma will be isolated from a portion of each subject's peripheral blood and bone marrow aspirate samples in an on-site laboratory. Each subject's de-identified LC gene sequence and their de-identified plasma samples will then be sent to Memorial Sloan-Kettering Cancer Center (MSKCC) for mass spectrometry to look for fragmentary protein sequences associated with the culprit LC gene of each subject.

After reaching a CR or VGPR, at annual evaluations for up to 3 years, the genomic DNA from the research sample of bone marrow collected during standard of care clinical procedures will be used to confirm maintenance of response by testing for the presence of MRD with each of the 3 methods (Q-PCR, WGS, and plasma protein analysis) noted above. Marrow material collected for the purposes of this study will not be stored after analysis, and primer-probe set design will be conducted entirely within Tufts Medical Center. Any marrow samples not fully consumed during analysis will be destroyed.

By using these three methods this protocol will determine whether one method is superior to the others and whether the three methods produce results that correlate with each other. The decision to discontinue participation in MRD testing will be made by the patient and the physician on an individual basis. Patients who have relapse or hematologic progression of disease during the three year period by standard blood and urine tests will no longer have testing for MRD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AL amyloidosis at Tufts Medical Center who have baseline bone marrow samples available and achieve a CR or VGPR to treatment. Patients may consent and register at diagnosis and have a baseline marrow collected at the time of consent; or patients may consent during therapy prior to achieving a response, if they have previously banked marrow cells for research.

Exclusion Criteria:

* Patients who do not have available baseline bone marrow samples.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will enroll AL amyloidosis patients at Tufts Medical Center who have baseline bone marrow cells available from the time of diagnosis, or from a time of therapy prior to achieving a response, and then subsequently achieve a CR or VGPR with first-line therapy. Up to 50 patients diagnosed with AL amyloidosis will be evaluated on this protocol.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2015-08; Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Minimal Residual Disease Testing by Q-PCR, NGS, and mass spectrometry | 3 years
  After achievement of a CR or VGPR, minimal residual disease testing (using Q-PCR, WGS, and plasma protein analysis by mass spectrometry) will be done annually for up to 3 years. These tests will show either the presence of absence of minimal residual disease. These findings will then be correlated with progression free survival as assessed through standard clinical tests for AL amyloidosis.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Comenzo, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Abraham RS, Geyer SM, Price-Troska TL, Allmer C, Kyle RA, Gertz MA, Fonseca R. Immunoglobulin light chain variable (V) region genes influence clinical presentation and outcome in light chain-associated amyloidosis (AL). Blood. 2003 May 15;101(10):3801-8. doi: 10.1182/blood-2002-09-2707. Epub 2002 Dec 19. PMID 12515719
- [Background] Perfetti V, Casarini S, Palladini G, Vignarelli MC, Klersy C, Diegoli M, Ascari E, Merlini G. Analysis of V(lambda)-J(lambda) expression in plasma cells from primary (AL) amyloidosis and normal bone marrow identifies 3r (lambdaIII) as a new amyloid-associated germline gene segment. Blood. 2002 Aug 1;100(3):948-53. doi: 10.1182/blood-2002-01-0114. PMID 12130507
- [Background] Bodi K, Prokaeva T, Spencer B, Eberhard M, Connors LH, Seldin DC. AL-Base: a visual platform analysis tool for the study of amyloidogenic immunoglobulin light chain sequences. Amyloid. 2009 Mar;16(1):1-8. doi: 10.1080/13506120802676781. PMID 19291508
- [Background] Comenzo RL. Plasma cell neoplasms, their precursor States, and their prediction of organ damage. J Clin Oncol. 2014 Sep 1;32(25):2679-82. doi: 10.1200/JCO.2014.56.2892. Epub 2014 Jul 14. No abstract available. PMID 25024079
- [Background] Comenzo RL, Wally J, Kica G, Murray J, Ericsson T, Skinner M, Zhang Y. Clonal immunoglobulin light chain variable region germline gene use in AL amyloidosis: association with dominant amyloid-related organ involvement and survival after stem cell transplantation. Br J Haematol. 1999 Sep;106(3):744-51. doi: 10.1046/j.1365-2141.1999.01591.x. PMID 10468868
- [Background] Comenzo RL, Zhang Y, Martinez C, Osman K, Herrera GA. The tropism of organ involvement in primary systemic amyloidosis: contributions of Ig V(L) germ line gene use and clonal plasma cell burden. Blood. 2001 Aug 1;98(3):714-20. doi: 10.1182/blood.v98.3.714. PMID 11468171
- [Background] Dasari S, Theis JD, Vrana JA, Meureta OM, Quint PS, Muppa P, Zenka RM, Tschumper RC, Jelinek DF, Davila JI, Sarangi V, Kurtin PJ, Dogan A. Proteomic detection of immunoglobulin light chain variable region peptides from amyloidosis patient biopsies. J Proteome Res. 2015 Apr 3;14(4):1957-67. doi: 10.1021/acs.jproteome.5b00015. Epub 2015 Mar 20. PMID 25734799
- [Background] van der Velden VH, Cazzaniga G, Schrauder A, Hancock J, Bader P, Panzer-Grumayer ER, Flohr T, Sutton R, Cave H, Madsen HO, Cayuela JM, Trka J, Eckert C, Foroni L, Zur Stadt U, Beldjord K, Raff T, van der Schoot CE, van Dongen JJ; European Study Group on MRD detection in ALL (ESG-MRD-ALL). Analysis of minimal residual disease by Ig/TCR gene rearrangements: guidelines for interpretation of real-time quantitative PCR data. Leukemia. 2007 Apr;21(4):604-11. doi: 10.1038/sj.leu.2404586. Epub 2007 Feb 8. PMID 17287850
- [Background] Wang Q, Xia J, Jia P, Pao W, Zhao Z. Application of next generation sequencing to human gene fusion detection: computational tools, features and perspectives. Brief Bioinform. 2013 Jul;14(4):506-19. doi: 10.1093/bib/bbs044. Epub 2012 Aug 9. PMID 22877769
- [Background] Welschof M, Terness P, Kolbinger F, Zewe M, Dubel S, Dorsam H, Hain C, Finger M, Jung M, Moldenhauer G, et al. Amino acid sequence based PCR primers for amplification of rearranged human heavy and light chain immunoglobulin variable region genes. J Immunol Methods. 1995 Feb 27;179(2):203-14. doi: 10.1016/0022-1759(94)00286-6. PMID 7876568
- [Background] Zhou P, Comenzo RL, Olshen AB, Bonvini E, Koenig S, Maslak PG, Fleisher M, Hoffman J, Jhanwar S, Young JW, Nimer SD, Boruchov AM. CD32B is highly expressed on clonal plasma cells from patients with systemic light-chain amyloidosis and provides a target for monoclonal antibody-based therapy. Blood. 2008 Apr 1;111(7):3403-6. doi: 10.1182/blood-2007-11-125526. Epub 2008 Jan 23. PMID 18216299
- [Background] Zhou P, Hoffman J, Landau H, Hassoun H, Iyer L, Comenzo RL. Clonal plasma cell pathophysiology and clinical features of disease are linked to clonal plasma cell expression of cyclin D1 in systemic light-chain amyloidosis. Clin Lymphoma Myeloma Leuk. 2012 Feb;12(1):49-58. doi: 10.1016/j.clml.2011.09.217. Epub 2011 Nov 18. PMID 22100494
- [Background] Zhou P, Ma X, Iyer L, Chaulagain C, Comenzo RL. One siRNA pool targeting the lambda constant region stops lambda light-chain production and causes terminal endoplasmic reticulum stress. Blood. 2014 May 29;123(22):3440-51. doi: 10.1182/blood-2013-10-535187. Epub 2014 Apr 10. PMID 24723680
- [Background] Zhao M, Wang Q, Wang Q, Jia P, Zhao Z. Computational tools for copy number variation (CNV) detection using next-generation sequencing data: features and perspectives. BMC Bioinformatics. 2013;14 Suppl 11(Suppl 11):S1. doi: 10.1186/1471-2105-14-S11-S1. Epub 2013 Sep 13. PMID 24564169
- [Background] Zhou P, Zhang Y, Martinez C, Kalakonda N, Nimer SD, Comenzo RL. Melphalan-mobilized blood stem cell components contain minimal clonotypic myeloma cell contamination. Blood. 2003 Jul 15;102(2):477-9. doi: 10.1182/blood-2002-12-3674. Epub 2003 Mar 20. PMID 12649134